CLINICAL TRIAL: NCT04390087
Title: Effect of Wheelchair-modified Upper-body Rowing Exercise on Traditional and Novel Cardiometabolic Risk Factors in Spinal Cord Injured Wheelchair Users - Protocol for a Randomized Controlled Trial
Brief Title: Effect of Upper-body Rowing on Cardiometabolic Risk in Spinal Cord Injured Wheelchair Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Aage og Johanne Louis-Hansens Fond (Other)
Responsible Party: Principal Investigator, Rasmus Kopp Hansen, Principal Investigator, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: N-20190053
Record Dates: First submitted 2020-05-06; First posted 2020-05-15 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Spinal Cord Injuries; Exercise Training
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Upper-body rowing performed up to 30 min, 3 times per week with moderate-to-vigorous intensity
  Interventions: Other: Exercise
- Control (No Intervention): The participants allocated to the control group will be asked to maintain their normal lifestyle throughout the intervention period

INTERVENTIONS:
Other: Exercise — Upper-body rowing performed while participants are sitting in their own wheelchair.
  Arms: Exercise

SUMMARY:
This randomized controlled trial will determine the effects of 12-weeks of wheelchair user-modified upper-body rowing on both traditional cardiometabolic risk factors in SCI manual wheelchair users.

DETAILED DESCRIPTION:
This randomized controlled trial aims to determine the effects of 12-weeks of wheelchair user-modified upper-body rowing on both traditional (insulin resistance, obesity, dyslipidemia (including low HDL-C and elevated TG and blood pressure) and novel (inflammatory status, autonomic nervous system function, vascular structure and function, and cardiorespiratory fitness level) cardiometabolic risk factors in SCI manual wheelchair users. As secondary objectives, this trial will investigate the effects of the exercise intervention on free-living physical activity, shoulder pain, and indices of quality of life.

Men and women, aged 18-65 years; chronic SCI (≥1 year since injury); individuals with sufficient sparing of arm function to participate in upper-body rowing; using a manual wheelchair as a primary tool for mobility will be included in the trial.

The exercise training will be conducted as wheelchair-modified upper-body ergometer rowing. The training will be performed for up to 30 min, 3 times per week with moderate-to-vigorous intensity, with at least one rest day between sessions.

Outcome measurements will be performed immediately before (baseline), after (post) 12 weeks of training, and 6 months after the termination of the intervention period (follow up). This approach allows for assessment of the short term effects of exercise training as well as any residual effects from the training intervention on cardiometabolic risk, shoulder pain, indices of quality of life, and free-living physical activity

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years;
* chronic SCI (≥1 year since injury)
* individuals with sufficient sparing of arm function to participate in upper-body rowing (i.e. as a minimum excluding individuals with complete SCI at or above C5)
* using a manual wheelchair as a primary tool for mobility.

Exclusion Criteria:

* Individuals who regularly engage in >150 min/week of moderate-to-vigorous intensity physical activity
* have received a cortisone injection in the shoulder within the last four months
* have had shoulder injury within the previous year
* known medical issues (urinary tract infections, cardiovascular contraindications for exercise testing, and pressure sores)
* diagnosed diabetes or any endocrine, heart, kidney, liver disease or any other disease that may limit the ability to perform exercise.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
fasting insulin | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  Serum fasting insulin concentration will be measured from approximately 20 mL blood drawn from a peripheral vein

SECONDARY OUTCOMES:
Arterial blood pressure | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  Resting systolic and diastolic BP will be measured with an automated blood pressure monitoring device
Body mass | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  Body mass (kg)
Heart rate variability (HRV) | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  HRV will be derived from spectral analysis of the R-R interval obtained from the ECG.
Vascular structure | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  Intima media thickness (mm)
Fasting blood glucose | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  Venous blood sampling
Cardiorespiratory fitness level | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  Peak oxygen consumption
Shoulder pain | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  the Wheelchair Users Shoulder Pain Index (WUSPI)). Consist of 15 items each consisting og a visual analog scales (pain from 0-10, with 10 representing maximum pain).
Free-living physical activity | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  Wrist-worn accelerometer
Health-related quality of life (HRQOL) | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  Short-form 36 (SF-36). 0-100, with 100 representing the best possible health.
body mass index | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  BMI (kg/m2)
Waist Circumference | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  Measured in cm
Conduit artery function | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  Flow-mediated dilation (percent change from baseline)
Resistance vessel function | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  Reactive hyperemia (blood flow area under the curve)
Vascular function | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  Blood flow (ml/min)
Long-term blood glucose | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  HbA1c (percent)
HDL cholesterol | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  Concentration (mmol/l)
LDL cholesterol | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  concentration (mmol/l)
Triglyceride | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  concentration (mmol/l)
C-reactive protein | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  mg/l
Alanin-aminotransferase | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  U/L
Interleukin 6 | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  Anti and pro-inflammatory cytokine
Tumor necrosis factor-alpha | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  Pro-inflammatory cytokine
Interleukin-10 | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  Antoinflammatory cytokine
Interleukin-1 receptor antagonist | The between group difference in change in outcome will be examined from baseline to post intervention (12-weeks follow-up) (primary endpoint) and again from 12-weeks follow-up to 6-months follow-up (secondary endpoint)
  Anti-inflammatory cytokine

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus K Hansen, MSc, Principal Investigator — Aalborg University
Locations (1):
- Aalborg University, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hansen RK, Laessoe U, Samani A, Mellergaard M, Rasmussen RW, Handberg A, Larsen RG. Impact of upper-body ergometer rowing exercise on aerobic fitness and cardiometabolic disease risk in individuals with spinal cord injury: A 6-month follow-up study. J Spinal Cord Med. 2024 Nov;47(6):996-1006. doi: 10.1080/10790268.2023.2233820. Epub 2023 Aug 3. PMID 37534922
- [Derived] Hansen RK, de Wit JLJ, Samani A, Laessoe U, Figlewski K, Larsen RG. Wheelchair-modified ergometer rowing exercise in individuals with spinal cord injury: a feasibility, acceptability, and preliminary efficacy study. Spinal Cord Ser Cases. 2022 Apr 30;8(1):48. doi: 10.1038/s41394-022-00518-6. PMID 35487894
- [Derived] Hansen RK, Samani A, Laessoe U, Handberg A, Larsen RG. Effect of wheelchair-modified rowing exercise on cardiometabolic risk factors in spinal cord injured wheelchair users: protocol for a randomised controlled trial. BMJ Open. 2020 Oct 16;10(10):e040727. doi: 10.1136/bmjopen-2020-040727. PMID 33067301